CLINICAL TRIAL: NCT03120156
Title: Effects of Sensomotoric Insoles on Postural Control in Elderly People - a Prospective Randomized Controlled Trial
Brief Title: Effects of Sensomotoric Insoles on Postural Control in Elderly People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, PD Dr. Martin Weigl, MPH, Principal investigator, Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Senso-Insoles for Balance
Record Dates: First submitted 2017-03-30; First posted 2017-04-19 (Actual); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Sensorimotor Gait Disorder
Keywords: sensomotoric insoles; postural control; proprioceptive insoles; insoles
MeSH Terms: conditions — Gait Disorders, Neurologic

STUDY DESIGN:
Intervention Model Description: Prospective randomized controlled trial
Masking Description: Sensomotoric insoles and normal insoles or no insoles are not maskable.Patients and all involved persons will be able to easily see which type of insoles are used.
  No blinding possible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No insoles (Active Comparator): Control group of people with poor postural control that won't use insoles
  Interventions: Other: No insoles
- Normal insoles (Active Comparator): Control group of people with poor postural control that will get normal standard insoles.
  Interventions: Device: normal standard insoles
- Sensomotoric insoles (Active Comparator): Control group of people with poor postural control that will get normal standard insoles.
  Interventions: Device: sensomotoric insoles

INTERVENTIONS:
Device: sensomotoric insoles — sensomotoric insoles were published by Jahrling (2007) and have a certain shape that could improve balance abilities. The toes 2-4 are higher that toe 1, so that the tendons of the toe-flectors are pre-stressed.
  Arms: Sensomotoric insoles
Device: normal standard insoles — Normal standard insole like you will get them by receipe from an orthotic shop
  Arms: Normal insoles
Other: No insoles — control group with no insoles in the shoes
  Arms: No insoles

SUMMARY:
People with weak balance ability or subjective feeling of dizziness and unsure gait are separated into 3 training-groups. One Group is getting no insoles, the second group is getting modern sensomotoric insoles, and the third group is getting normal standard insoles. All are passing a 6 week proprioceptive training.

Main outcome measurements are posturography at baseline, 3 weeks and 6 weeks. Secondary measurements are ABC-Scale, Tinetti Gait and balance test and functional reach test at baseline and after 6 weeks.

DETAILED DESCRIPTION:
People with weak balance ability or subjective feeling of dizziness and unsure gait are separated into 3 training-groups. Exclusion criteria are structural neuropathic cause for dizziness, severe ocular deficience, cochlear causes for dizziness.

The 3 Groups differ in following criteria:

Group 1: Gets basic insoles after 3-D-Scan of the foot Group 2: Gets sensomotoric insoles (Jahrling) after 3-D-Scan of the foot. Group 3: Control-Group = no insoles

Alle groups are doing a 6 weeks proprioceptive training 2 times a week for 45min. Balance-Ability is measured by a posturographic plate prior to the training, after 3 weeks training and after 6 weeks of training. ABC-Score, Tinetti Gait and Balance test and functional reach test are secondary outcome measurements and are evaluated prior the training and after 6 weeks of training.

ELIGIBILITY:
Inclusion Criteria:

ABC-Scale < 70% Functional reach test < 30cm Subjective feeling of unsure gait or several falls in the last 5 years

Exclusion Criteria:

Structural pathologies in the balance system Neuropathologies like Polyneuropathy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2017-10-27 (Actual); Study Completion 2017-10-27 (Actual)

PRIMARY OUTCOMES:
Posturographic measurement with Kistler's measuring plate | 30 min.
  a validated posturgraphy plate is measuring the balance ability

SECONDARY OUTCOMES:
Tinetti Balance and Gait instrument | 15 min.
  Well established tool for measuring balance ability of elderly people
Functional reach test | 5 min
  Well established tool for measuring balance ability
ABC-Scale | 15 min
  Questionnaire-Score for evaluation subjective feelings of unsure gait patterns or dizziness

CONTACTS AND LOCATIONS:
Locations (1):
- Ludwig Maximilian University, University Hosipital, Department of Orthopedics, Physical Medicine and Rehabilitation, Munich, Germany

IPD SHARING:
Plan to Share IPD: No